CLINICAL TRIAL: NCT03138434
Title: Advanced MRI in AAA
Status: Terminated | Type: Observational
Why Stopped: Sufficient acquisitions for DCE-MRI and 4D flow, but not for T1/T2-mapping due to lack of ILT in some participants.
Sponsor: Ron Balm (Other)
Responsible Party: Sponsor-Investigator, Ron Balm, prof. dr., Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Organization: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Other Study IDs: NL56823.018.16
Record Dates: First submitted 2017-05-01; First posted 2017-05-03 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Abdominal Aortic Aneurysm
Keywords: Abdominal Aortic Aneurysm; 4D flow MRI; DCE-MRI; T1 and T2 mapping
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Optimization phase: The first five patients will be included for the optimization of the MRI sequences. This is to ensure that a standard protocol will work for different sizes of AAA. These patients will only be scanned once.
- Study phase: This phase will commence after the optimization phase. This phase is where we want to assess the feasibility, reproducibility and association with disease severity between MRI parameters and AAA.
  These twenty patients will be scanned twice, with an interval of 1 week ± 5 days.
  The study will be completed when we have 20 patients with 2 scans for each sequence, or when a maximum number of 30 patients in the study phase have been scanned.

SUMMARY:
This study aims to determine whether advanced MRI sequences can provide robust and clinically relevant information about abdominal aortic aneurysms (AAAs). The MRI sequences will study outcomes related to blood flow inside AAA, microvasculature of the AAA vessel wall and intraluminal thrombus inside AAA.

Robustness of these MRI sequences will be determined with testing of feasibility and reproducibility. Clinical relevance will be assessed by studying the association between the primary outcomes and disease severity. Disease severity will be expressed by AAA diameter.

It is our hypothesis that these parameters are significantly related to disease severity and may therefore be future markers of disease progression.

DETAILED DESCRIPTION:
This prospective study evaluates the feasibility, reproducibility and clinical relevance of MRI sequences in adults with an abdominal aortic aneurysm (AAA).

The MRI sequences and their primary outcomes are:

* Four-dimensional (4D) flow MRI and wall shear stress (WSS)
* Dynamic Contrast-Enhanced (DCE) MRI and kinetic transport constant (Ktrans)
* T1 and T2 mapping (T1 and T2 relaxation times)

Feasibility is tested by the production of high-quality images that enable calculation of the primary outcomes. Reproducibility is tested by calculating interscan, intra- and interobserver variability. Clinical relevance is tested by assessing the association between primary outcomes and disease severity which is expressed by AAA diameter

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥ 18 years of age)
* Abdominal aortic aneurysm with a maximal aneurysm diameter of at least 30 mm

Exclusion Criteria:

* Contra-indications for MRI
* Severely reduced renal function (eGFR < 30)
* Previous allergic reaction to intravenous contrast agents
* Suprarenal AAA
* Pararenal AAA
* Previous aneurysm repair
* Inflammatory aneurysm
* Mycotic or other infectious aneurysm
* Vasculitis
* Connective tissue disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with an abdominal aortic aneurysms who are patients at the department of vascular surgery of the Academic Medical Center.
Sampling Method: Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2017-04-12 (Actual); Primary Completion 2019-05-29 (Actual); Study Completion 2019-05-29 (Actual)

PRIMARY OUTCOMES:
Wall shear stress (WSS) | Time of MRI scan
  Primary outcome of 4D flow MRI
Kinetic transport constant (Ktrans) | Time of MRI scan
  Primary outcome of DCE-MRI
T1 relaxation time | Time of MRI scan
  Primary outcome of T1 mapping
T2 relaxation time | Time of MRI scan
  Primary outcome of T2 mapping

SECONDARY OUTCOMES:
Peak flow velocity inside the aneurysm | Time of MRI scan
  Secondary outcome of 4D flow MRI
Location of peak wall shear stress | Time of MRI scan
  Secondary outcome of 4D flow MRI
Flow velocity at aneurysm entrance | Time of MRI scan
  Secondary outcome of 4D flow MRI
Flow patterns | Time of MRI scan
  Secondary outcome of 4D flow MRI
Oscillatory shear index | Time of MRI scan
  Secondary outcome of 4D flow MRI
Reverse reflux rate constant (kep) | Time of MRI scan
  Secondary outcome of DCE-MRI
Area under the curve of contrast uptake | Time of MRI scan
  Secondary outcome of DCE-MRI
Peak enhancement ratio | Time of MRI scan
  Secondary outcome of DCE-MRI
Wash-in slope | Time of MRI scan
  Secondary outcome of DCE-MRI
Time to peak (TTP) | Time of MRI scan
  Secondary outcome of DCE-MRI
Mean transit time (MTT) | Time of MRI scan
  Secondary outcome of DCE-MRI

CONTACTS AND LOCATIONS:
Overall Officials: Ron Balm, MD PhD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (1):
- Department of Vascular Surgery, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided